CLINICAL TRIAL: NCT03738787
Title: Efficacy and Safety of Exocrine Pancreatectomy With Neoprene®-Based Glue After High-risk Pancreatoduodenectomy (PD) in Patients With Pancreatic, Papilla, Duodenal, and Distal Choledochus Neoplasm
Brief Title: Treatment of the Pancreatic Stump With Neoprene®-Based Glue After High-risk Pancreatoduodenectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Vincenzo Mazzaferro, Professor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191/14
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Fistula; Pancreatic Neoplasms; Postoperative Complications
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms; Postoperative Complications | interventions — Neoprene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreatic duct occlusion (Experimental): Patients considered at high risk for pancreatic fistula or oncological relapse due to introperative evaluation submitted to pancreatic duct occlusion with Neoprene-based glue.
  Interventions: Procedure: Pancreatic duct occlusion with Neoprene
- Pancreato-Jejunal anastomosi (Active Comparator): Patients considered at low risk for pancreatic fistula submitted to pancreato-jejunal anastomosis.
  Interventions: Procedure: Pancreato-Jejunal anastomosis

INTERVENTIONS:
Procedure: Pancreatic duct occlusion with Neoprene — Pancreatic duct occlusion of the pancreatic stump with Neoprene-based glue after Pancreatoduodenectomy.
  Arms: Pancreatic duct occlusion
Procedure: Pancreato-Jejunal anastomosis — Standardized pancreato-jejunal anastomosis after Pancreatoduodenectomy
  Arms: Pancreato-Jejunal anastomosi

SUMMARY:
The study evaluates the safety and efficacy of Neoprene-based glue in the management of pancreatic stump after pancreatoduodenectomy (PD) in patients at high risk for pancreatic fistula and early neoplastic recurrence, compared with a population of patients at conventional risk.

DETAILED DESCRIPTION:
Although improved in many aspects, the PD intervention is still burdened by a significant morbidity, related above all to the delicate phase following the removal of the tumor which involves the reconstruction of the gastro-enteric, biliary and especially pancreatic pathway. Among the many variants of the reconstructive phase, that of pancreato-jejunal anastomosis is the one burdened by the highest complication rate (quantified around 40%, with a percentage of pancreatic fistula between 5% and 35%).

In cases at risk of pancreatic fistula it is possible not to perform a conventional pancreato-jejunal anastomosis, but to decide to inject into the pancreatic stump the solidifying glues with the aim of inducing a chemical pancreatectomy of the exocrine component of the pancreas.

Neoprene® (Polychloroprene) has the property of polymerizing and solidifying in an environment with a pH lower than its own (pH <12).

After a systematic review of the sporadic experiences of chemical pancreatectomy published until today, due to the increased complexity of the surgical cases of patients undergoing PD, the investigators have undertaken a formal, single-center prospective study, aimed at clarifying the safety and efficacy data of a Neoprene®-based glue in patients selected through objective criteria (such as the high risk of pancreatic fistula and early tumor recovery after pancreatoduodenectomy).

In this study is expected the prospective collection of a cohort of patients with tumor of the head of the pancreas, papilla, duodenum and distal choledochus to undergo pancreatoduodenectomy (PD) at high risk of pancreatic fistula and / or local recurrence ("Study Arm").

At the same time a second cohort of patients with the same type of neoplasia will be collected, subjected to PD intervention in which however it will be possible to proceed with pancreato-jejunal anastomosis. This group will be defined as "Control Arm".

The first cohort will be the group of patients in which to detect the safety and efficacy of the treatment with Neoprene®-based glue.

The second cohort will be the comparative control group against which patients treated with Neoprene®-based glue can be compared in the hypothesis that peri-operative morbidity,mortality and short and long-term side effects of the intervention are equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an alternative-Fistula Risk Score >15%.
* Patients with insulin-dependent diabetes.
* Cirrhotic patients or with histologically proven chronic liver disease.
* Age> 75 years (relative criterion, ie insufficient by itself to justify the procedure and therefore to be associated with one of the other cited criteria).
* Patients with intraoperative demonstration on histological examination of lymph node metastasis;
* Patients with R1 interventions.
* Presence of minimal extra-pancreatic tumor disease not detected pre-operatively (nodule of carcinosis, single liver metastasis) and removed with the primary tumor within the same intervention;
* Patients undergoing preoperative radiotherapy / chemotherapy for tumors reconverted to surgical operability.

Exclusion Criteria:

* All other patients who undergo PD in which the eligibility conditions for the study group are not present, are enrolled in the Control Arm..

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative complications of grade > II according to Dindo-Clavien classification | 90 days
  Comparison of 90-days clinically relevant postoperative morbidity rate of grade > II according to Dindo-Clavien classification between the two arms.
Rate of overall postoperative complications | 90 days
  Comparison of 90-days overall postoperative morbidity rate of any grade according to Dindo-Clavien classification between the two arms.
Rate of postoperative mortality | 90 days
  Comparison of 90-days postoperative mortality rate between the two arms

SECONDARY OUTCOMES:
Number of participants with onset of post-surgical diabetes | 12 months
  Comparison between arms of onset of newly diagnosed post-surgical diabetes needing tablets or insulin therapy during a follow-up period of 12 months
Percentual variation of weight after pancreatoduodenectomy | 12 months
  Comparison between arms of percentual weight variation between preoperative measure in kilograms and follow up at 1, 3, 6 and 12 months
Variation of Body Mass Index after pancreatoduodenectomy | 12 months
  Comparison between arms of Body Mass Index variation measured combining weight and height to report BMI in kg/m^2 between preoperative evaluation and follow up at 1, 3, 6 and 12 months

OTHER OUTCOMES:
Overall survival | 36 months
  Evaluation of overall survival in both arms of study

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazzaferro V, Virdis M, Sposito C, Cotsoglou C, Droz Dit Busset M, Bongini M, Flores M, Prinzi N, Coppa J. Permanent Pancreatic Duct Occlusion With Neoprene-based Glue Injection After Pancreatoduodenectomy at High Risk of Pancreatic Fistula: A Prospective Clinical Study. Ann Surg. 2019 Nov;270(5):791-798. doi: 10.1097/SLA.0000000000003514. PMID 31567180